CLINICAL TRIAL: NCT03380910
Title: An Interprofessional Intervention With Behavioral Health and Pharmacy Trainees to Reduce Smoking Rates at a Free Health Clinic in Richmond
Brief Title: An Interprofessional Intervention to Reduce Smoking Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20010390
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Smoking, Cigarette
MeSH Terms: conditions — Cigarette Smoking | interventions — Dosage Forms; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ready to Quit (Experimental): Current patients who speak Spanish, smoke cigarettes, and are ready to quit will be included. The intervention includes an interdisciplinary team approach using pharmacy and behavioral health trainees to provide smoking cessation services.
  Interventions: Behavioral: Pharmacy and Behavioral Health Team
- Not Ready to Quit (Other): Current patients who speak Spanish, smoke cigarettes, and are not ready to quit will be included. The intervention includes an interdisciplinary team approach using pharmacy and behavioral health trainees to provide smoking cessation services.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Pharmacy and Behavioral Health Team — An interdisciplinary approach using medications through pharmacy support and counseling through behavioral health team members will be used to improve smoking cessation rates.
  Arms: Ready to Quit
Behavioral: Motivational Interviewing — Patients not ready to quit will be offered motivational interviewing to increase readiness to quit.
  Arms: Not Ready to Quit

SUMMARY:
The purpose of this study is to test the effectiveness of an experimental process to aid Spanish-speaking patients in quitting smoking with the help of pharmacists and behavioral health psychologist trainees and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Spanish-speaking
* Uninsured
* Current cigarette smoker

Exclusion Criteria:

* Pregnant or breastfeeding
* Heart attack or stroke in the last 3 months

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Change in smoking abstinence | Baseline to 6 months
  Smoking abstinence will be measured by breath carbon monoxide level

SECONDARY OUTCOMES:
Change in Readiness to Quit Smoking | Baseline to 6 months
  Improvement in readiness to quit will be measured by the quit ladder
Change in Nicotine Dependence | Baseline to 6 months
  Nicotine dependence will be measured by the Fagerstrom scale
Change in Number of Cigarettes Smoked | Baseline to 6 months
  Change in the number of cigarettes smoked will be measured by patient reported values
Change Carbon Monoxide Levels | Baseline to 6 months
  Measured by Carbon Monoxide Meter

CONTACTS AND LOCATIONS:
Locations (1):
- CrossOver Healthcare Ministry, Henrico, Virginia, United States